CLINICAL TRIAL: NCT06426394
Title: The Effect of End-expiratory Positive Pressure on Gastric Residual Volume in Elective Pediatric Outpatient Surgery Where Laryngeal Mask is Applied
Brief Title: Effect of Positive End-expiratory Pressure on Gastic Residual Volume
Status: Completed | Type: Observational
Sponsor: Duygu Akyol (Other Government)
Collaborators: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Duygu Akyol, M.D, co-investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Organization: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Other Study IDs: 2023-541
Record Dates: First submitted 2024-05-14; First posted 2024-05-23 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pediatrics; Fasting Period
Keywords: Gastric ultrasonography; gastric residual volume; pediatric outpatient surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study was designed as a prospective observational study.

DETAILED DESCRIPTION:
In this study, it was planned to evaluate the effect of positive end-expiratory pressure on gastric residual volume in patients who will undergo outpatient pediatric surgery with laryngeal mask application on the specified dates. Patients aged 1-11 years, ASA I-II and undergoing outpatient lower abdominal and genitourinary surgery were included in the study. Since the use of positive end-expiratory pressure varies in our clinic depending on the anesthesiologist preference, the effect of this application on gastric volume will also be evaluated primarily by recording images with gastric ultrasonography at certain perioperative time periods. Secondarily, the effect of this positive end-expiratory pressure on mechanical ventilator parameters and airway pressures will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients who will undergo elective outpatient minor surgery (lower abdominal and urogenital)
* 1-11 years old
* American Society of Anesthesiology (ASA) classification 1-2 patient groups
* Patients who are fully hungry and whose fasting period is appropriate for their age and diet.

Exclusion Criteria:

* Patients whose fasting period is not appropriate
* Acute abdominal and emergency surgeries
* ASA 3-4 patient group
* Patients with diseases or medication use that will affect gastric emptying time
* Previous nasogastric tube placement and re-operation • Patients with known difficult airway or failure to fit the laryngeal mask

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A total of 90 patients were planned for this study.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-05-17 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Gastric residual volume | preoperatively, intraoperatively after laryngeal mask placement, before laryngeal mask removal at the end of surgery
  The primary purpose of this study is to measure gastric residual volume with peroperative gastric ultrasonography measurements. Gastric residual volume will be calculated according to gastric ultrasonography measurements.

SECONDARY OUTCOMES:
Airway pressures | intraoperative process
  The secondary aim of this study was to evaluate the effect of positive end-expiratory pressures on airway pressures

CONTACTS AND LOCATIONS:
Locations (1):
- Duygu Akyol, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gunasekaran A, Govindaraj K, Gupta SL, Vinayagam S, Mishra SK. Comparison of Gastric Insufflation Volume Between Ambu AuraGain and ProSeal Laryngeal Mask Airway Using Ultrasonography in Patients Undergoing General Anesthesia: A Randomized Controlled Trial. Cureus. 2022 Aug 11;14(8):e27888. doi: 10.7759/cureus.27888. eCollection 2022 Aug. PMID 36110490
- [Background] Sharma G, Jacob R, Mahankali S, Ravindra MN. Preoperative assessment of gastric contents and volume using bedside ultrasound in adult patients: A prospective, observational, correlation study. Indian J Anaesth. 2018 Oct;62(10):753-758. doi: 10.4103/ija.IJA_147_18. PMID 30443057
- [Background] Beck CE, Rudolp D, Becke-Jakob K, Schindler E, Etspuler A, Trapp A, Fink G, Muller-Lobeck L, Roher K, Genahr A, Eich C, Sumpelmann R. Real fasting times and incidence of pulmonary aspiration in children: Results of a German prospective multicenter observational study. Paediatr Anaesth. 2019 Oct;29(10):1040-1045. doi: 10.1111/pan.13725. Epub 2019 Sep 4. PMID 31435997
- [Background] Fiedler MO, Schatzle E, Contzen M, Gernoth C, Weiss C, Walter T, Viergutz T, Kalenka A. Evaluation of Different Positive End-Expiratory Pressures Using Supreme Airway Laryngeal Mask during Minor Surgical Procedures in Children. Medicina (Kaunas). 2020 Oct 21;56(10):551. doi: 10.3390/medicina56100551. PMID 33096743